CLINICAL TRIAL: NCT03811938
Title: Catheter ABlation of Low Voltage Regions in the Treatment of Persistent Atrial Fibrillation (ABLOVO-AF Study)
Brief Title: Ablation of Low Voltage Regions in Persistent Atrial Fibrillation
Acronym: ABLOVO-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS 202816
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Radiofrequency Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Vein Isolation (Active Comparator): Historical control from cases performed in year 2017 at Hammersmith Hospital. Intervention: Pulmonary vein isolation.
  Interventions: Procedure: Pulmonary Vein Isolation
- Low voltage ablation (Experimental): Active arm, Intervention: Standard pulmonary vein isolation and Low Voltage Ablation.
  Interventions: Procedure: Low voltage ablation

INTERVENTIONS:
Procedure: Low voltage ablation — Catheter ablation of low voltage areas in the left atrium and catheter ablation aiming for the electrical isolation of the pulmonary veins.
  Arms: Low voltage ablation
Procedure: Pulmonary Vein Isolation — Catheter ablation aiming for the electrical isolation of the pulmonary veins.
  Arms: Pulmonary Vein Isolation

SUMMARY:
Background. Atrial fibrillation (AF) is a disorganised rhythm of the upper chambers of the heart. It can lead to severe complications including stroke or heart failure. It can be treated with radiofrequency ablation (RFA). This technology works by heating heart muscle inside the heart to break the electrical circuits responsible for the abnormal rhythm.

The energy is delivered into the heart with plastic tubes that have metal electrodes, inserted through the groin veins and removed after the procedure. The patient is usually put to sleep during the intervention.

If the AF has been present for more than seven days but for less than one year it is called persistent, and it can be difficult to treat successfully with the usual methods.

Goals. The study will test a new RFA technique to treat patients with persistent AF. This involves identifying areas within the left upper chamber that have a lower electrical voltage than the surrounding heart muscle and applying RFA to the border zones of these areas.

Methods. The new technology combined with the usual procedure will be compared to the usual procedure alone. All patients will receive ablation according to the new technique and results will be compared to a historical control group from the trial institution.

Follow up. Patients will be followed up for 12 months with clinic visits and heart rhythm checks.

Potential benefit. The new technique will be assessed for success at keeping patients free from persistent AF compared to the usual methods.

The study will be performed at Imperial College Healthcare NHS Trust, at the Hammersmith Hospital. Licensed clinical software will be used from St Jude Medical to guide ablation and a special research software module will be used to analyse data from the heart following ablation. The study will be sponsored by Imperial College Healthcare NHS Trust

ELIGIBILITY:
Inclusion Criteria:

1. Suitable candidate for catheter mapping/ablation for arrhythmias.
2. Eighteen (18) to eighty-five (85) years of age
3. Body Mass Index (BMI) < 40 (Wt. in Kgs / Ht. in m2)
4. Signed Informed Consent

Exclusion Criteria:

1. Severe cerebrovascular disease
2. Moderate to severe renal impairment (eGFR < 30)
3. Active gastrointestinal bleeding
4. Active infection or fever
5. Short life expectancy
6. Significant anemia
7. Severe uncontrolled systemic hypertension
8. Severe electrolyte imbalance
9. Ejection fraction of < 35%
10. Congestive heart failure (NYHA Class IV)
11. Unstable angina requiring emergent PTCA (percutaneous transluminal coronary angioplasty) or CABG (coronary artery bypass graft)
12. Recent myocardial infarction
13. Bleeding or clotting disorders
14. Uncontrolled diabetes
15. Inability to receive IV or oral Anticoagulants
16. Unable to give informed consent (these patients would not be recruited)
17. Previous catheter or surgical ablation treatment for atrial fibrillation.
18. Paroxysmal atrial fibrillation.
19. Pregnancy (urinary pregnancy test will be offered on the day of the procedure for all women of reproductive age)
20. Drug and/or alcohol abuse
21. Transient factors for AF
22. Severe LA enlargement of >60 mm in diameter on echocardiography
23. Patients who have participated in another study of an investigational medicinal product in the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 3-12 months.
  Recurrence of atrial arrhythmia of at least 30s in duration. Investigation period for arrhythmia recurrence will be between 3 and 12 months after the first procedure, allowing for a blanking period of 3 months.

SECONDARY OUTCOMES:
Canadian Cardiovascular Society Severity in Atrial Fibrillation Score | 12 months
  Canadian Cardiovascular Society Severity in Atrial Fibrillation (CCS-SAF) change.
  0 represents no symptoms, 4 represents symptoms that significantly interfere with quality of life and exercise capacity.
Antiarrhythmic drugs | 3-12 months
  Change in the number of antiarrhythmic drugs per patient
Number of AF ablations | 3-12 months
  Number of additional AF ablations
Complication rate | 3-12 months
  Number and rate of complications in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Phang B Lim, MB BChir, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No